CLINICAL TRIAL: NCT06215365
Title: Study of Health-risk Behaviours (Tobacco, Alcohol or Drug Consumption ; Nutrition ; Sedentary Lifestyle ; Sexual Practices) Among Cancer Survivors
Acronym: PREVAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL23_1306
Record Dates: First submitted 2023-12-27; First posted 2024-01-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Cancer Remission
Keywords: Health-risk behaviours; post-cancer; prevention; screening; vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult cancer survivors (until 74 years old) who have completed their heavy treatments (Experimental): Adult cancer survivors (until 74 years old) who have completed their heavy treatments (chemotherapy, radio-chemotherapy, …) and that are taking part in the "JUMP post-cancer day" which is a multidisciplinary evaluation carried out at the end of treatments.
  They must not have cognitive disorders that limit their ability to understand and complete the questionnaire. Also, they have to speak, read and write French language.
  The study will be presented to the patient who can refuse to participate. The digital version of the questionnaire will be handed out, if the patient does not object after a period of thinking, when he or she comes to the day hospital for his or her JUMP Day. The study will therefore take place at a single point in time, and no pre-inclusion or follow-up visits are planned as part of this protocol.
  Completing the questionnaire takes about 15 to 20 minutes. All questions are designed to meet the stated objectives. No personally identifiable data is collected.
  Interventions: Behavioral: Adult cancer survivors who have completed their heavy treatments

INTERVENTIONS:
Behavioral: Adult cancer survivors who have completed their heavy treatments — The study will be presented to the patient who can refuse to participate. The digital version of the questionnaire will be handed out, if the patient does not object after a period of thinking, when he or she comes to the day hospital for his or her JUMP Day. The study will therefore take place at a single point in time, and no pre-inclusion or follow-up visits are planned as part of this protocol.
  Completing the questionnaire takes about 15 to 20 minutes. All questions are designed to meet the stated objectives. No personally identifiable data is collected.

SUMMARY:
* Cancer is now becoming a chronic condition though it was, until a short time ago, a fatal illness. Thus, according to the French national cancer institute, nearly 4 million French people have been diagnosed with cancer in their lifetime.
* Screening is used to detect the presence of a pathology at an early, infra-clinical stage, or the presence of a risk factor in people who are supposedly healthy.
* There are three organized screening programs in France (breast cancer, colorectal cancer, cervical cancer), as well as many others recommended by learned societies such as the National Authority for Health . However, they are underused, far from European recommendations and government targets.
* According to DREES (research, studies, evaluation and statistic department), public health and primary prevention interventions could have prevented 143 deaths per 100.000 inhabitants, and healthcare interventions could have spared 59 deaths per 100.000 inhabitants, for a total of 202 avoidable deaths per 100.000 inhabitants in France in 2020.
* As for cancers, French national cancer institute estimates the rate of avoidable cancers in France in 2023 at 40%. Breast cancer, for example, is the most common cancer that can be associated with alcohol consumption and estimations suggest that nearly 20.000 breast cancers could be prevented each year (a third of new cancer cases in 2018).
* In France, prevention accounts for 5.5% of healthcare expenses in 2021, with 46% for individual primary prevention, 41% for individual secondary prevention and 12% for collective prevention and prevention programs. These healthcare expenses must be set against the social cost of each risk factor, to see how important they are.
* Relative burden of cancer and noncancer mortality among long-term survivors of breast, prostate, and colorectal cancer in the US has been demonstrated. It shows that "patients with low oncologic risk at the time of diagnosis had at least 3-fold higher risk of noncancer death compared with death from the index cancer".
* In France, medical desertification is a reality. Now, according to the VICAN-5 study, nearly a third of cancer patients are not followed up by general practitioners. Though primary prevention is one of GP's prerogatives and a governmental priority.
* There is a high interest in screening and preventive action to limit the risk of other avoidable pathologies, whether cancerous or not.

The research hypothesis is that a customized screening will enable the implementation of comprehensive preventive action to limit the onset of avoidable diseases (second cancer or other pathology) for cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivor
* Up to 74 years old
* Less than a year from the end of their heavy treatments
* Participating in JUMP post-cancer day.

Exclusion Criteria:

* Patients with cognitive disorders that limit their ability to understand and complete the questionnaire.
* Patients who do not speak, read and write French.

Ages: 74 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
The percentage of people in the studied population with at least one modifiable health risk behavior among cancer survivors. | through study completion, an average of 2 months
  Modifiable health risk behaviors are: tobacco, alcohol or drug consumption ; nutrition ; sedentary lifestyle ; sexual practices.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] STOLTZ Justine. Mise en place d'une intervention d'évaluation des comportements à risques et de dépistage dans l'après-cancer (CO5). Congrès PARKOURS onco-hémato 2025, Auditorium Pasteur, jeudi 30 janvier 2025, 17:45-18:00 (Lyon).